CLINICAL TRIAL: NCT02466178
Title: Multicenter Efficacy Trial of the Serene RF System for the Reduction of Glabellar Lines
Brief Title: Efficacy Trial for the Reduction of Glabellar Lines
Status: Completed | Type: Observational
Sponsor: Serene Medical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SM 14-01
Record Dates: First submitted 2015-03-11; First posted 2015-06-09 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Rhytids in the Glabellar Region

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Serene RF System: Percutaneous delivery of radiofrequency (RF) energy to create a temporary conduction block to the corrugator and/or procerus muscles.
  Interventions: Device: Serene RF System

INTERVENTIONS:
Device: Serene RF System — The Serene RF System provides percutaneous delivery of radiofrequency (RF) energy to a targeted nerve.

SUMMARY:
The purpose of this study is to evaluate the ability of the Serene RF System to effectively improve the appearance of dynamic glabellar lines and sustain the effect for a minimum of 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Glabellar lines rating of at least two per the Merz Scale
2. Written informed consent
3. Understands and accepts the following obligations during the follow-up period (minimum of three months and up to one year)
4. available for the 3 day phone call and present for each follow-up visit;
5. receive NO other facial procedures in the upper face for a minimum of three months and up to one year after the RF procedure;
6. make NO changes to the eyebrows for a minimum of three months after the RF procedure.

Exclusion Criteria:

1. Injection of botulinum toxin to the upper face within the previous four months
2. Use of fillers in the upper face within the previous twelve months
3. Use of prescription treatments (e.g., Renova, Retin-A, micro-dermabrasion, chemical peels) on the upper face, in the area between the eyebrows where frown lines occur, within the previous four weeks or plans to use these treatments during the study
4. Facial or skin conditions that could interfere with treatment or confound results (e.g., signs or symptoms of eyebrow or eyelid ptosis, facial nerve palsy, scarring, infection)
5. Implanted pacemaker or automatic implantable cardioverter/defibrillator
6. History of keloid formation
7. Known bleeding disorder
8. Use of thrombolytics, anticoagulants, aspirin or non-steroidal anti-inflammatory drugs within seven days prior to study treatment Is receiving systemic corticosteroids or anabolic steroids (standard doses of inhaled or nasal corticosteroids are acceptable)
9. History of chronic or recurrent infection, or compromised immune system
10. Known lidocaine hypersensitivity
11. Enrollment in another research study
12. Pregnant, or plans to get pregnant during the follow-up period
13. Any other condition or circumstance that might either pose a risk, in the investigator's opinion, to the subject or interfere with the ability to acquire satisfactory clinical data throughout the follow-up period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult men and women with moderate to severe glabellar lines
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The reduction of glabellar lines | 3 months
  The reduction of glabellar lines will be assessed by a panel of 3 independent reviewers with expertise in dermatology and/or plastic surgery of the change in glabellar lines measured from baseline to 3, 6, 9 and 12 months post procedure. Photographs will be presented in a random order and the reviewers will be blinded to whether the photograph is baseline or a follow up. Effectiveness of the procedure is defined by a ≥ 1 point improvement in score (i.e., numerical decrease) on the Mertz Aesthetics Scale™ (Merz Scale) for dynamic glabellar lines. At each time point the severity of the glabellar lines is assessed on a 5 point scale.

SECONDARY OUTCOMES:
Incidence and severity of adverse events | 3 months
The reduction of glabellar lines | 12 months
  The reduction of glabellar lines will be assessed by a panel of 3 independent reviewers with expertise in dermatology and/or plastic surgery of the change in glabellar lines measured from baseline to 3, 6, 9 and 12 months post procedure. Photographs will be presented in a random order and the reviewers will be blinded to whether the photograph is baseline or a follow up. Effectiveness of the procedure is defined by a ≥ 1 point improvement in score (i.e., numerical decrease) on the Mertz Aesthetics Scale™ (Merz Scale) for dynamic glabellar lines. At each time point the severity of the glabellar lines is assessed on a 5 point scale.
Subject satisfaction | 12 months
  Subject satisfaction will be assessed by a survey given every 3 months. This survey asks the subject questions to rate on a scale of 0-4 with 0 representing very dissatisfied and 4 representing very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Scott McGill, Study Director — Vice President Product Development
Locations (5):
- United States (5):
  - Premier Plastic Surgery, Palo Alto, California
  - Premier Plastic Surgery, San Mateo, California
  - Aesthetic Plastic Surgery, New York, New York
  - Reviance Plastic Surgery & Aesthetics Center, Clackamas, Oregon
  - Puget Sound Plastic Surgery, Kirkland, Washington